CLINICAL TRIAL: NCT05938855
Title: Prospective Evaluation of the Performance and Safety of PHENIX LIBERTY, a Medical Device for Electrostimulation and Biofeedback, in the Treatment of Pelvic Static Disorders in Women With Urinary Incontinence.
Brief Title: Performance and Safety of the PHENIX LIBERTY, a Medical Device for Electrostimulation and Biofeedback, in the Treatment of Pelvic Static Disorders in Women With Urinary Incontinence.
Acronym: IncontiLib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivaltis (Industry)
Collaborators: CEISO (Industry); Human Physio (Unknown); Pôle santé de la Nartassière (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A02195-40
Record Dates: First submitted 2023-06-22; First posted 2023-07-11 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Urinary Incontinence; Pelvic Floor Disorders
Keywords: Electrical stimulation; Biofeedback
MeSH Terms: conditions — Urinary Incontinence; Pelvic Floor Disorders | interventions — Electric Stimulation; Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard of care plus additional questionaire (Other): As part of this clinical investigation, the medical device under investigation is used in accordance with its usual use, and the patient's therapeutic procedure includes additional, non-invasive procedures. These additional procedures relate to the addition of an end-of-life visit and validated questionnaires assessing functional deficiencies and impact on daily life.
  Interventions: Device: Electrical stimulation and biofeedback with the medical device Phenix Liberty

INTERVENTIONS:
Device: Electrical stimulation and biofeedback with the medical device Phenix Liberty — The patient will undergo 10 therapeutic functional re-education sessions, at regular intervals according to a schedule drawn up by the physiotherapist, during which the PHENIX LIBERTY device may be used.
  The patients will complete questionnaires at the end of the care Overall, the functional perineal rehabilitation sessions will include muscle testing, electrostimulation and biofeedback.
  The follow up will be conduct as follow :
  * 10 sessions between 10 and 12 weeks
  * 1 end visit, within the week after the 10th session

SUMMARY:
The goal of this clinical trial is to evaluate the short-term improvement in urinary incontinence after perineo-sphincter rehabilitation using functional electrostimulation and biofeedback (PHENIX LIBERTY VIVALTIS device) in patients with pelvic statics disorders.

• Does the use of the medical device in the treatment of pelvic static disorders lead to an improvement in urinary incontinence?

Participants will use the medical device, which provides electrical stimulation, biofeedback and pressure biofeedback to re-educate the pelvic floor muscles and improve urinary incontinence.

DETAILED DESCRIPTION:
Rational :

Urinary incontinence is a condition affecting many women in their adult lives. It is considered a public health problem, and has a high negative impact on patients' quality of life. Physiotherapy-based perineal rehabilitation is considered the first-line treatment for this condition. Treatments consist of pelvic floor muscle exercises (physiotherapy) with or without the use of other resources such as biofeedback, electrical electro-stimulation and vaginal cones.

In this context, the promoter wishes to carry out this study in order to reinforce the data currently available on the medical device PHENIX LIBERTY.

Design:

Prospective, interventional with non invasive and non burdensome procedure, non-comparative, multicenter, open-label study of a CE-marked medical device.

Intervention :

As part of this clinical investigation, the medical device under investigation is used in accordance with its usual use, and the patient's therapeutic procedure includes additional, non-invasive procedures. These additional procedures relate to the addition of an end-of-life visit and validated questionnaires assessing functional deficiencies and impact on daily life.

The care will be conduct as follow:

* 1 inclusion visit (V0) (from 1 say to 15 days prior the the first functional therapeutic re-education session)
* 10 sessions of functional therapeutic re-education, during which the PHENIX LIBERTY device may be used. Sessions performed at regular intervals according to a schedule drawn up by the physiotherapist (between 10 and 12 weeks)
* 1 end visit (V11), 1 week after the 10th session to complet questionnaires

In total, the patient will be followed 15 weeks maximum

ELIGIBILITY:
Inclusion Criteria:

* Patient who is incontinent (involuntary loss of urine) and/or has an overactive bladder (pollakiuria defined as more than one nocturnal urination and more than six daytime urination or leakage per day); Incontinent patient requiring functional rehabilitation of pelvic static disorders by electrostimulation and biofeedback;
* Adult patient (between 18 / 75 years old);
* Patient with at least one of the following symptoms related to a pelvic static disorder: pain, hypertonia, muscle weakness, decreased or loss of motor control, trophic abnormality;
* Patient who can make herself available to participate in the sessions regularly and who believes that she will be able to complete the tenth treatment session no later than 8 weeks after V0;
* Patient who has signed the consent form to participate in the study;
* Patient physically and mentally willing and able, in the judgment of the investigator at the time of recruitment, to perform the procedures under study;
* Patient with social protection.

Exclusion Criteria:

* Patient with peripheral or central neurological involvement (perianal or perivulvar sensitivity disorder);
* Patient with BMI ≥30 kg/m²
* Patient who has had more than 3 deliveries;
* Patient with stroke, Alzheimer's, multiple sclerosis, spinal cord involvement, narrow lumbar canal, cauda equina syndrome, or cognitive and/or behavioral impairment that may, in the practitioner's judgment, interact with the self-questionnaire or biofeedback assessment;
* Pregnant woman at the inclusion visit;
* Patient with an implanted pacemaker or spinal cord trainer;
* Patient with hypersensitivity to electrostimulation;
* Patient with such vaginal atrophy that an endovaginal probe cannot be used
* Patient with chronic or recurrent vaginal or urinary tract infection on long-term treatment;
* Patient with vaginal pathology (undiagnosed bleeding, cancer in the area to be treated);
* Patient who has renounced her liberty by administrative or judicial sentence, or who is under guardianship or limited judicial protection;
* Patient participating in an interventional clinical trial or testing/having tested an investigational drug and/or medical device within 30 days prior to inclusion in the study in relation to the relevant pathology;
* Patient who cannot read or write French;
* Patient refusing to participate in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Changes in the frequency of bladder weakness | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  A mictional grid will be used
  The mictional grid covers a period of forty-eight to seventy-two hours. It assesses the number of micturitions during the day and at night, and quantifies the volume of urine passed at each micturition, as well as diuresis over a 24-hour period. The mictional grid visualizes episodes of leakage, their quantity (small drops, beginning of micturition or massive leakage) and the moment of onset, such as during effort (coughing, sneezing, carrying a load, sport, etc.) or at rest.

SECONDARY OUTCOMES:
Changes in the Pelvic Floor Impact Questionnaire (PFIQ-7) score assessing the impact of pelvic static disorders | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  The Pelvic Floor Impact Questionnaire (PFIQ-7) will be used, it assess the social impact of pelvic statics disorders.
  The questionnaire has 7 questions and 3 columns. The first column concerns urinary symptoms, the 2nd column concerns colorectal-anal symptoms and the 3rd column concerns genital prolapse symptoms.
  All questions use the following answer format:
  * Not at all = 0
  * Somewhat = 1
  * Moderately = 2
  * A lot = 3
  Each column gives a score between 0 and 100, which will be added to give the total score of the PFIQ-7 scale between 0 and 300.
  A high score indicates a significant impact of pelvic static disorders
Change in patients' visual analog scale (VAS) pain scores | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  The pain caused by the pelvic floor disorder will be assessed by the Visual Analogue Scale (VAS).
  The VAS is made up of a 10-centimeter line anchored by two ends of the pain. 10 is the first end being the "maximum pain imaginable" and 0 is the other end being "no pain".
Changes in the number of voids during the day and at night, | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  The number of voids during the day and at night will be assessed.
  The same mictional grid will be used
  The mictional grid covers a period of forty-eight to seventy-two hours. It assesses the number of micturitions during the day and at night, and quantifies the volume of urine passed at each micturition, as well as diuresis over a 24-hour period. The mictional grid visualizes episodes of leakage, their quantity (small drops, beginning of micturition or massive leakage) and the moment of onset, such as during effort (coughing, sneezing, carrying a load, sport, etc.) or at rest.
Change in the severity of leakage | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  The severity of leakage will be assessed (small drops, onset of micturition or massive leakage)
  The same mictional grid will be used
  The mictional grid covers a period of forty-eight to seventy-two hours. It assesses the number of micturitions during the day and at night, and quantifies the volume of urine passed at each micturition, as well as diuresis over a 24-hour period. The mictional grid visualizes episodes of leakage, their quantity (small drops, beginning of micturition or massive leakage) and the moment of onset, such as during effort (coughing, sneezing, carrying a load, sport, etc.) or at rest.
Change in diuresis over twenty-four hours; | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  The number of voiding sensation over twenty-four hours will be assessed
  The same mictional grid will be used
  The mictional grid covers a period of forty-eight to seventy-two hours. It assesses the number of micturitions during the day and at night, and quantifies the volume of urine passed at each micturition, as well as diuresis over a 24-hour period. The mictional grid visualizes episodes of leakage, their quantity (small drops, beginning of micturition or massive leakage) and the moment of onset, such as during effort (coughing, sneezing, carrying a load, sport, etc.) or at rest.
Change in the volume of urine voided at each voiding | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  The volume of urine voided at each voiding will be assessed in deciliter
  The same mictional grid will be used
  The mictional grid covers a period of forty-eight to seventy-two hours. It assesses the number of micturitions during the day and at night, and quantifies the volume of urine passed at each micturition, as well as diuresis over a 24-hour period. The mictional grid visualizes episodes of leakage, their quantity (small drops, beginning of micturition or massive leakage) and the moment of onset, such as during effort (coughing, sneezing, carrying a load, sport, etc.) or at rest.
Changes in the rate of improvement in perineal protection reflex during a coughing effort | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  A surface Electromyography (EMG) will be used. Muscle electrical activity provides a "map" of muscle recruitment according to exercise conditions (position, relative load, type of resistance, type of support, etc.).
Changes in the rate of improvement of hypertonia assessed through measurement of myoelectric activity | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  A surface Electromyography (EMG) will be used. Muscle electrical activity provides a "map" of muscle recruitment according to exercise conditions (position, relative load, type of resistance, type of support, etc.).
Changes in the rate of improvement in hypertonia assessed through measurement of perineal muscle tone | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  Modified Oxford gradient will be used. This is an assessment of pelvic floor muscle strength by the practitioner, using vaginal palpation.
  The score is scored as follows: 0 → no detectable pelvic floor contraction , 1 → very weak pelvic floor contraction, 2 → weak pelvic floor contraction, 3 → moderate pelvic floor contraction, 4 → good pelvic floor contraction, 5 → strong pelvic floor contraction
Evolution of vaginal microcirculation and trophicity according to the practitioner's subjective opinion | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  This outcome will be assessed according to the practitioner's opinion regarding visual assessment, palpation assessment of the vagina.
  The practitioners will indicated if on his opinion there is a an abnormal vaginal microcirculation and trophicity.
Changes in the rate of improvement in awakening and muscle strengthening assessed through measurement of myoelectric activity | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  A surface Electromyography (EMG) and a vaginal intra-cavity probe will be used. Muscle electrical activity provides a "map" of muscle recruitment according to exercise conditions (position, relative load, type of resistance, type of support, etc.).
Changes in the rate of improvement in awakening and muscle strengthening assessed through measurement of perineal muscle tone | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  Modified Oxford gradient will be used. This is an assessment of pelvic floor muscle strength by the practitioner, using vaginal palpation.
  The score is scored as follows: 0 → no detectable pelvic floor contraction , 1 → very weak pelvic floor contraction, 2 → weak pelvic floor contraction, 3 → moderate pelvic floor contraction, 4 → good pelvic floor contraction, 5 → strong pelvic floor contraction
Percentage of patients with an improvement in pelvic statics | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  This outcome will be assessed according to the practitioner's opinion
Incidence of adverse events | At each visit, from day 0 to Week 15 (at the end visit within the week after the 10th seance)
  Rate of the incidence of adverse events related to the medical device
Evaluation of the Global Impression of Change Scale score after therapeutic management | Week 15 (at the end visit within the week after the 10th seance)
  The Patient's Global Impression of Change (PGIC) Scale is a questionnaire designed to express the patient's overall impression of changes in symptoms, activities, emotions and quality of life following therapeutic treatment17. The patient answers the first question by ticking one of the proposed answers, each answer corresponding to a score from 1 to 7. The patient then scores his or her impression of progress on a scale from 0 to 10.
Evaluation of responses to the patient satisfaction questionnaire on the use of the PHENIX LIBERTY device after therapeutic management | Week 15 (at the end visit within the week after the 10th seance)
  The satisfaction questionnaire is constructed on the basis of the Likert Scale. The sponsor has written an questionnaire regarding the use of the Phenix Liberty for the patient.
  The Likert scale (or attitude scale) is a semantic rating system, generally consisting of 5 or 7 items, used in surveys to measure and evaluate perceptions, attitudes and opinions.
  The evaluation will be based on the following responses: Strongly agree (=5) ; Agree (=4) ; Rather agree (=3) ; Rather disagree (=2) ; Disagree (=1= ; Strongly disagree (=0).
  The minimum score 0 means a worse outcome and the maximum score 5 means a better outcome.
Evolution of the vaginal lubrication and hydration score for the evaluation of microcirculation and vaginal trophicity | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  Vaginal lubrication and hydration can also be used to assess vaginal microcirculation and trophicity. This parameter is observed by the practitioner through visual and tactile observation. The score is as follows: 1 → no vaginal lubrication/hydration (altered mucosa), 2 → no vaginal lubrication/hydration (unaltered mucosa), 3 → very low vaginal lubrication/hydration, 4 → moderate vaginal lubrication/hydration, 5 → normal vaginal lubrication/hydration.
Evolution of the vaginal acidity score for assessing vaginal microcirculation and trophicity | Day 0 and Week 15 (at the end visit within the week after the 10th seance)
  Vaginal pH is an important element in determining vaginal health, encompassing microcirculation and vaginal trophicity. The vagina is an acidic environment (pH ≤ 4.6) thanks to its healthy bacterial flora, which secrete lactic acid to limit the growth of many pathogenic microbes. A scale will be used to frame the different pH values. The score is as follows: 1 → pH ≥6.1, 2 → pH = 5.6-6, 3 → 5.1-5.5, 4 → 4.7-5.0, 5 → ≤4.6. (Appendix 6bis) Score 1 represents an abnormal pH and score 5 represents a normal pH.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Willame, Principal Investigator — Human Physio; Julie Perrin, Principal Investigator — Pôle santé de la Nartassière
Locations (2):
- France (2):
  - Pôle santé de la Nartassière, Mouans-Sartoux
  - Human Physio, Nîmes